CLINICAL TRIAL: NCT05057962
Title: Tocilizumab for Treatment of SARS Cov2 Pneumonia. Experience in a Private Health Center Facility in Buenos Aires City.
Brief Title: Tocilizumab in Covid-19 Penumonia in Buenos Aires City
Status: Completed | Type: Observational
Sponsor: Sanatorio Finochietto (Other)
Responsible Party: Principal Investigator, Nazareno Galvalisi, Doctor, Sanatorio Finochietto
Other Study IDs: 5489
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Pneumonia; Tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We conducted a retrospective observational study of adult participants receiving only SOC (dexamethasone 8 mg or its equivalent plus oxygen, HNFO or eventual IMV) versus participants receiving SOC plus TCZ (8mg/kg as a single dose) as treatment for severe or critical SARS CoV2 pneumonia. The inclusion date will be the date of admission, and follow up will conclude at death or discharge (whichever occurs first) to describe clinical and laboratory characteristics and outcome of adult participants receiving only standard of care (SOC) versus participants receiving SOC plus TCZ as treatment for severe or critical SARS CoV2 pneumonia.

DETAILED DESCRIPTION:
Settings Emergency Department, General Ward and Intensive Care Unit (ICU) at Sanatorio Finochietto in Buenos Aires City, Argentina. Sanatorio Finochietto is a third level health care facility that provides health care services in prevalent clinical and surgical pathologies. It has the formerly mentioned units; as well as a Maternity Ward and complementary services (such as Laboratory, Radiology and Hemodynamics) and a total of 161 beds 30 of which are ICU beds.

Population Adult participants 18 years old and older receiving SOC plus TCZ versus only SOC as treatment for severe or critical SARS CoV2 pneumonia in Sanatorio Finochietto, between March 1st and August 31st 2021.

Participants in the control group couldn't receive TCZ because they were out of therapeutic window or had secondary infections suspicion.

Exposure variable is TCZ yes/no.

Inclusion Criteria

* Participants 18 years and older at admission.
* Confirmed diagnosis of severe SARS CoV 2 infection.
* Participants in category 6 and 7 of World's Health Organization (WHO) COVID 19 ordinal scale on Clinical Improvement (in Annexa).

Variables of study

Sociodemographics:

Sex. Categoric, dichotomous. M: male. F: female. Age. At time of admission. Numerical, continual, in years. Weight. At time of admission. Numerical, continual, in kg. Height. Numerical, continual, in cm. Body Mass Index (BMI). Numerical, continual. It will be calculated by the formula weight/height2.

Clinical characteristics Medical History. Nominal category. 1: Asthma 2: Chronic Obstructive Pulmonary Disease (COPD) 3: Diabetes (DBT) 4: High blood pressure (HBP) 5: Obesity 6: Coronary disease 7: Heart failure 8: Solid Tumor 9: Oncohematologycal diseasse 10: Person living with Human Immunodeficiency Virus (PLWHIV).

Acute Physiology and Chronic Health Evaluation II (APACHE II). Numerical, continual.

Symptoms onset date. Numerical, continual. Admission date. Numerical, continual. Steroids onset date. Numerical, continual. Total steroids days. Numerical, continual. Defined as dexamethasone dose equal or over 8 mg.

Methylprednisolone pulse. Nominal category. Yes/No. Defined as infusion of at least 500 mg methylprednisolone.

Number of methylprednisolone pulses. Numerical, continual. IMV. Nominal category. Yes/No. IMV days. Numerical, continual. HNFO. Nominal category. Yes/No. HFNO. Numerical, continual. Shock. Nominal category. Yes/No. Defined as vasopressor requirements for 24 hours or more.

Other organ failure. Nominal category. Yes/No. Defined as organ failure besides hemodinamic or respiratory failure.

Worsening date. Numerical, continual. Worsening is defined as more oxygen requirement (non rebreather mask or high nasal flow oxygen).

TCZ infusion. Nominal category. Yes/no. TCZ infusion date. Numerical, continual. TCZ dose. Numerical, continual. TCZ adverse reaction. Nominal category. Yes/No. Defined as adverse reaction during infusion, neutropenia at 24/48 hs and 7th day or discharge (whichever occurs first) and/or hepatic enzymes elevation above five times normal value at 24/48 hs and 7th day or discharge (whichever occurs first).

WHO COVID 19 ordinal scale on Clinical Improvement at worsening. Numerical, continual.

WHO COVID 19 ordinal scale on Clinical Improvement at 14th day or discharge (whichever occurs first). Numerical, continual.

CRP value. Numerical, continual. At tociluzumab's infusion date or closest previous.

Ferritin value. Numerical, continual. At tociluzumab's infusion date or closest previous.

D dimer value. Numerical, continual. At tociluzumab's infusion date or closest previous.

CRP value at discharge. Numerical, continual. At discharge or closest previous. Ferritin value at discharge. Numerical, continual. At discharge or closest previous.

D dimer value at discharge. Numerical, continual. At dishcarge or closest previous.

Secondary infections. Open Survival. Nominal category. Yes/no. Cause of death. Open. Discharge date. Numerical, continual.

Data circuit Information will be collected from electronic records. Given that all severe SARS CoV 2 pneumonia participants with SOC or SOC plus TCZ will be included, sample calculation won't be estimated.

Statistical analysis In the descriptive analysis, quantitative data are expressed as mean and standard deviation or median and interquartile range 25-75 (IQR) according to their distribution. Data normality was evaluated using charts and Kolmogorov-Smirnov's test. Qualitative data are expressed as absolute and relative frequency in percentage. For comparison between groups, chi2 or Fisher test were used according to assumptions for qualitative data and Wilcoxon for quantitative data according to their distribution. A significance level of less than 0.05 was considered. R software version 4.0.3 was used.

Ethical considerations This investigation will be conducted under national and international regulatory rules about human health investigations; and according to Ministry Resolutions, Helsinki declaration and all its amendments and Good Clinical Practice Guidelines ICH E6.

All study data will be processed with the utmost confidentiality and anonymously, with restricted access only to authorized personnel and for study purposes only according to current legislation of National Personal Data Protection Laws (Ley de Habeas data) and Law 26529/09.

Data will be encoded using a numerical code randomly generated. This code will replace the patient's name and last name. Identificatory data in database comprehensed in the 18 identifiers of HIPPA rules will be eliminated (A su vez se eliminarán los datos identificatorios de la base de datos a analizar comprendido por los 18 identificadores detallados por las normas HIPAA). Database will be saved in a computer and accessed with a code and only by the principal investigator. After statistical analysis it will be eliminated.

This is an observational study and uses a secondary database, and constitutes a minimal risk investigation; so according to CIOMS 2016 and Pauta 10, exception of informed consent for participants is requested.

Endpoints Secondary infections, death at discharge, WHO COVID 19 ordinal scale on Clinical Improvement at 14 days from worsening or discharge (whichever occurs first).

Financing Cost in administrative and human resources for the study will be assumed by principal investigators. There will be no extraordinary costs for subjects nor health care providers.

Interest conflicts Investigators declares none interest conflicts

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older at admission.
* Confirmed diagnosis of severe SARS CoV 2 infection.
* category 6 and 7 of World's Health Organization (WHO) COVID 19 ordinal scale on Clinical Improvement .

Exclusion Criteria:

under 18 years of age no Confirmed diagnosis of SARS CoV 2 infection. category 1dnd 5 of World's Health Organization (WHO) COVID 19 ordinal scale on Clinical Improvement .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants 18 years old and older receiving SOC plus TCZ versus only SOC as treatment for severe or critical SARS CoV2 pneumonia in Sanatorio Finochietto, between March 1st and August 31st 2021.
  Participants in the control group couldn't receive TCZ because they were out of therapeutic window or had secondary infections suspicion.
  Exposure variable is TCZ yes/no.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Death | From the date of admission to the date of death from any cause or discharge from hospital, whichever occurs first
  death during hospitalization
Secondary infections | From the date of admission to the date of death from any cause or discharge from hospital, whichever occurs first
  infection demonstrated with cultures of blood, urine, or respiratory specimens during hospitalization
WHO COVID 19 ordinal scale on Clinical Improvement and the 14 days | 14 days
  difference in the who ordinal scale between the date of worsening and the 14 days of the same, with 1 being the best value and 8 the worst (death)

CONTACTS AND LOCATIONS:
Locations (1):
- Nazareno Galvalisi, Buenos Aires, Argentina

DOCUMENTS (1):
  • Study Protocol (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT05057962/Prot_000.pdf